CLINICAL TRIAL: NCT05021146
Title: Essential Oil for Chronic Low Back Pain
Acronym: ECAP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Buda Health Center (Other)
Collaborators: dōTERRA International (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DO-221014-COP
Record Dates: First submitted 2021-08-18; First posted 2021-08-25 (Actual); Last update posted 2021-10-15 (Actual); Status verified 2021-10

CONDITIONS: Chronic Low-back Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Standard care and CEO treatment with standard 20% concentration Copaiba oil (Experimental)
  Interventions: Other: usual care and topical essential copaiba oil
- Standard care and CEO treatment with 40% concentration Copaiba oil (Experimental)
  Interventions: Other: usual care and topical essential copaiba oil
- standard care and placebo treatment with coconut oil (Placebo Comparator)
  Interventions: Other: usual care and placebo treatment
- Standard care (Active Comparator)
  Interventions: Other: usual care

INTERVENTIONS:
Other: usual care and topical essential copaiba oil — All subjects will receive daily interdisciplinary - multimodular -treatment during their hospital stay including a daily 30 minute massage therapy. Both experimental groups and the placebo group patients continue to use topical treatment in the first half of the follow up period (90 days).
  Arms: Standard care and CEO treatment with 40% concentration Copaiba oil; Standard care and CEO treatment with standard 20% concentration Copaiba oil
Other: usual care and placebo treatment — All subjects will receive daily interdisciplinary - multimodular -treatment during their hospital stay including a daily 30 minute massage therapy. Both experimental groups and the placebo group patients continue to use topical treatment in the first half of the follow up period (90 days).
  Arms: standard care and placebo treatment with coconut oil
Other: usual care — All subjects will receive daily interdisciplinary - multimodular -treatment during their hospital stay.
  Arms: Standard care

SUMMARY:
The specific objective of this study is to assess the safety and clinical efficacy of a new individualised spinal rehabilitation programme involving copaiba essential oil (CEO) therapy compared to usual care for people with chronic low back pain. Research in complementary and alternative medicine has increased over the last 15 years. As biochemical research shows, these substances carry the ability to relieve pain and to reduce inflammation. In doing so, it aims to:

1. Improve the health outcomes for individuals with chronic low back pain (CLBP) by positively impacting their pain, disability, work capacity, physical activity and mental health, and
2. Reduce the chronic health burden on society associated with treatment, sick leave, rehabilitation, and involuntary retirement, by reducing health-related costs.

The primary clinical hypothesis is that patients with CLBP receiving individualised spinal care and additional CEO topical treatment will have superior short- and long-term outcome (defined by condition specific quality of life and general well-being) compared to usual care.

ELIGIBILITY:
Inclusion Criteria:

* Chronic low back pain with or without irradiating pain (pain > 3 months)
* Low back pain is the dominant symptom, and Visual Analog Pain Scale (low back pain)>4
* Normal cognitive function, voluntary participation
* Able to read and answer the questionnaires in English or Hungarian language

Exclusion Criteria:

* Previous spinal surgery
* Untreated metabolic bone disease
* Active malignant disease
* Pregnancy
* Severe osteoporosis, fracture or posttraumatic deformity
* Spinal infection
* Neuromuscular disease
* Autoimmune disease
* Myelopathy
* Congenital spinal deformity
* Mental disorders
* Severe sciatica
* Severe spinal instability
* Refusing the study protocol

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2023-03-31 (Estimated); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | 6 months
  Visual Analogue Scale measured on a scale 0-10 where the higher the number the worse the pain intensity
Function | 6 months
  Oswestry Disability Index

SECONDARY OUTCOMES:
Core Outcome Measures Index Back (COMI Back) | 6 months
  A brief instrument for assessing the main outcomes of importance to patients with back problems (pain, function, symptom-specific well-being, quality of life, disability).
Quality of Life | 6 months
  EuroQoL-5D
Psychological measurements- Fear Avoidance Beliefs | 6 months
  Fear Avoidance Beliefs Questionnaire
Psychological measurements- Depression | 6 months
  Beck Depression Inventory
Psychological measurements- Pain catastrophization: | 6 months
  Pain Catastrophizing Scale
Psychological measurements- Anxiety | 6 months
  State-Trait Anxiety Inventory
Spinal function | 6 months
  Timed Up and Go (TUG) test
Spinal active range of motion | 6 months
  range of motion
Global treatment outcome | 6 months
  7- point Likert scale ( higher numbers representing worse the outcome)
Patient satisfaction | 6 months
  5- point Likert scale (smaller number represent more satisfied patients)
Demand of treatment | 6 months
  Pain medication and applied therapies after discharge

CONTACTS AND LOCATIONS:
Overall Officials: Peter Pal Varga, MD, Principal Investigator — Buda Health Center
Locations (1):
- National Center for Spinal Disorders / Buda Health Center, Budapest, Hungary

IPD SHARING:
Plan to Share IPD: No